CLINICAL TRIAL: NCT06106633
Title: Pain Reduction and Ovarian Perfusion Following Uterine Fibroid Embolization Via Pressure-Enabled Drug Delivery With the TriNav Infusion System (PEDD-UFE)
Brief Title: Pain Reduction and Ovarian Perfusion Following Uterine Fibroid Embolization
Acronym: PEDD-UFE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Principal Investigator, Dania Daye, MD, PhD, Assistant Professor of Radiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002406
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Uterine Bleeding; Uterine Fibroid
MeSH Terms: conditions — Uterine Hemorrhage; Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention Arm (Experimental): Patient will undergo UFE using PEDD
  Interventions: Device: TriNaV

INTERVENTIONS:
Device: TriNaV — Assess Pain Reduction and Ovarian Perfusion Following Uterine Fibroid Embolization Via Pressure-Enabled Drug Delivery With the TriNav Infusion System

SUMMARY:
The goal of this study is to assess of Pressure-Enabled Drug Delivery on fibroid treatment in patients undergoing UFE.

DETAILED DESCRIPTION:
Uterine fibroids are the most common tumor type in women of reproductive age and may be associated with abnormal menstrual bleeding, pain, sub-fertility, and diminished quality of life. For women interested in uterine preservation who want to derive adequate relief from medical management, uterine fibroid embolization (UFE) is a treatment option. The goal of this study is to assess of Pressure-Enabled Drug Delivery on fibroid treatment in patients undergoing UFE.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged >18 years.
2. Prior clinical decision for treatment by UFE.
3. One or more enhancing intramural, submucosal or subserosal fibroids on MRI.
4. Having either bulk symptoms or menorrhagia.

Exclusion Criteria:

1. Absolute contraindication to contrast-enhanced MRI.
2. Current pregnancy.
3. Known history of adenomyosis.
4. Diagnosis of pelvic inflammatory disease.
5. Diagnosis of endometriosis.
6. Post-menopausal (no menses >12-months).
7. Diagnosed gynecologic malignancy.
8. Prior uterine fibroid embolization treatment.
9. >50% volume of non-enhancing fibroids.
10. Prior oophorectomy
11. GnRH agonist therapy within 6-months or GnRH antagonist therapy within 1-month prior to entering the study.
12. Target uterine vasculature not suitable for treatment with the TriNav Infusion System.
13. Allergy or intolerance to dilaudid.
14. Lack of ovarian perfusion on baseline MRI.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | 6 months
  The Visual Analog Scale (VAS) Pain score will be used to assess pre- and post-procedural pain. The scale is from 1 to 10 with 1 indicating no pain and 10 indicating extreme pain.

SECONDARY OUTCOMES:
ovarian perfusion | 6 months
  Ultrasound doppler imaging will be used to assess changes in ovarian perfusion post-intervention compared to baseline ultrasound imaging

CONTACTS AND LOCATIONS:
Overall Officials: Dania Daye, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No